CLINICAL TRIAL: NCT01351948
Title: A Phase Ia Study to Assess the Safety and Immunogenicity of Novel Schedules for Vaccination With the Candidate Malaria Vaccines; AdCh63 AMA1, MVA AMA1 & AMA1-C1/Alhydrogel® +/- CPG 7909
Brief Title: Safety and Immunogenicity of Malaria Vaccines AdCh63 AMA1, MVA AMA1 and AMA1-C1/Alhydrogel®+/- CPG 7909
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC044
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Malaria
Keywords: Immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental): AdCh63 AMA1 + MVA AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909
  Interventions: Biological: AdCh63 AMA1 + MVA AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909
- Group 2 (Experimental): AdCh63 AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909
  Interventions: Biological: AdCh63 AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909
- Group 3 (Experimental): AdCh63 AMA1 + AMA1-C1/Alhydrogel®
  Interventions: Biological: AdCh63 AMA1 + AMA1-C1/Alhydrogel®
- Group 4 (Experimental): AdCh63 AMA1 AMA1-C1/Alhydrogel®+ CPG 7909
  Interventions: Biological: AdCh63 AMA1 AMA1-C1/Alhydrogel®+ CPG 7909
- Group 5 (Experimental): AdCh63 AMA1 + MVA AMA1
  Interventions: Biological: AdCh63 AMA1 + MVA AMA1

INTERVENTIONS:
Biological: AdCh63 AMA1 + MVA AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909 — 5x10^10 vp AdCh63 AMA1 Day 0, 1.25x10^8 pfu MVA AMA1 Day 56, AMA1-C1/Alhydrogel®+ CPG 7909 (80ug, 800ug, 564ug respectively) Day 112. IM injections
  Arms: Group 1
Biological: AdCh63 AMA1 + AMA1-C1/Alhydrogel®+ CPG 7909 — 5x10^10 vp AdCh63 AMA1 Day 0,AMA1-C1/Alhydrogel®+ CPG 7909 (80ug, 800ug, 564ug respectively) Day 56. IM injections
  Arms: Group 2
Biological: AdCh63 AMA1 + AMA1-C1/Alhydrogel® — 5x10^10 vp AdCh63 AMA1 Day 0, AMA1-C1/Alhydrogel® (80ug, 800ug respectively) Day 56. IM injections
  Arms: Group 3
Biological: AdCh63 AMA1 AMA1-C1/Alhydrogel®+ CPG 7909 — 5x10^10 vp AdCh63 AMA1 Day 0, AMA1-C1/Alhydrogel®+ CPG 7909 (80ug, 800ug, 564ug respectively) Day 112. IM injections
  Arms: Group 4
Biological: AdCh63 AMA1 + MVA AMA1 — 5x10^10 vp AdCh63 AMA1 Day 0, 1.25x10^8 pfu MVA AMA1 Day 112. IM injections
  Arms: Group 5

SUMMARY:
This study aims to compare the safety and immunogenicity of AdCh63 AMA1 and MVA AMA1vaccine candidates administered alone and with adjuvants in various schedules. These vaccines consist of inactivated viruses which have been modified, so they cannot reproduce in humans, and also to include genetic material for malaria protein AMA1 which is expressed by the malaria parasite during blood stage infection. The vaccines are designed to stimulate an immune response to this malaria protein and thus provide protection against malaria infection. Adjuvants are a crucial component of modern vaccine regimens, increasing the immunogenicity and potency of protein vaccines. In this study we will assess whether virus vectored vaccines combined with protein in adjuvant AMA1-C1/Alhydrogel® and CPG 7909 adjuvant (emulsion containing TLR agonist) can induce stronger and more durable immune response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* Women only: Must practice continuous effective contraception for the duration of the study.
* Men only: Must use barrier contraception from day of any vaccination with CPG 7909, for 3 months.
* Agreement to refrain from blood donation during the course of the study and for 6 months after the end of their involvement in the study.
* Written informed consent

Exclusion Criteria:

* History of clinical P. falciparum malaria
* Travel to a malaria endemic region during the study period or within the preceding six months with a significant risk of malaria exposure.
* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, lactation or intention to become pregnant during the study
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine e.g. egg products, Kathon.
* History of clinically significant contact dermatitis.
* History of a known allergy to nickel (volunteers may be enrolled in group 5 if they have an allergy to nickel)
* Any history of anaphylaxis post vaccination.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV).
* History or evidence of pre-existing autoimmune or antibody mediated disease or laboratory evidence of possible autoimmune disease, defined as anti-dsDNA ≥ 25 IU/mL or a positive antinuclear antibody (ANA) result at screening.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety of vaccination | Expected average of 12 months
  To assess the safety of vaccination of healthy adults with AdCh63 AMA1, MVA AMA1 & AMA1-C1/Alhydrogel® +/- CPG 7909 administered in various schedules using actively and passively collected data on adverse events

SECONDARY OUTCOMES:
Immunogenicity of vaccination | Expected average of 12 months
  To assess the immunogenicity of vaccination of healthy adults with AdCh63 AMA1, MVA AMA1 & AMA1-C1/Alhydrogel® +/- CPG 7909 administered in various schedules by measuring T cell responses (IFN-γ ELISPOT, flow cytometry), B cell responses and antibody responses to AMA1. Further immunological assessments may be undertaken as necessary

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil, FRCP, Principal Investigator — The Jenner Institute, University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Old Road, Headington, Oxford, United Kingdom